CLINICAL TRIAL: NCT02474641
Title: Adjuvant Radiotherapy After Breast-conserving Surgery in Early Breast Cancer: Hypofractionation With Simultaneous Integrated Boost vs. Standard Fractionation
Brief Title: Hypofractionation With Simultaneous Integrated Boost vs. Standard Fractionation in Early Breast Cancer
Acronym: HYPOSIB
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Schleswig-Holstein (Other)
Collaborators: University of Luebeck (Other)
Responsible Party: Principal Investigator, Juergen Dunst, Prof., Juergen Dunst, Prof., University Hospital Schleswig-Holstein
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARO-2013-05, ZKS-121-001
Record Dates: First submitted 2015-06-04; First posted 2015-06-18 (Estimated); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Early-Stage Breast Carcinoma
Keywords: Breast cancer; Hypofractionation with SIB; Non-inferiority; adjuvant radiotherapy with simultaneous integrated boost
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard radiation (Active Comparator): Conventionally fractionated radiotherapy of the breast followed by a tumor bed boost sequentially or
  Conventionally fractionated radiotherapy of the breast with simultaneous integrated boost to the tumor bed or
  Hypofractionated radiotherapy of the breast followed by a tumor bed boost sequentially
  Interventions: Radiation: Standard Radiation
- Hypofractionation with SIB (Experimental): Hypofractionated radiotherapy of the breast with simultaneous integrated boost to the tumor bed
  Interventions: Radiation: Hypofractionation with SIB

INTERVENTIONS:
Radiation: Standard Radiation — Conventionally fractionated radiotherapy of the breast followed by a tumor bed boost sequentially or
  Conventionally fractionated radiotherapy of the breast with simultaneous integrated boost to the tumor bed or
  Hypofractionated radiotherapy of the breast followed by a tumor bed boost sequentially
  Arms: Standard radiation
Radiation: Hypofractionation with SIB — Hypofractionated radiotherapy of the breast with simultaneous integrated boost to the tumor bed
  Arms: Hypofractionation with SIB

SUMMARY:
Hypofractionation with simultaneous integrated boost has been investigated in a few trials and appears to be safe and feasible.

Investigators initiated this multicenter two-armed phase III prospective trial to analyse the non-inferiority of hypofractionation with simultaneous integrated boost in patients with early breast cancer in comparison to standard fractionation.

DETAILED DESCRIPTION:
Control Arm:

Conventionaly fractionated radiotherapy of the breast 28 × 1.8 Gy = 50.4 Gy followed by a tumor bed boost sequentially 5 to 8 × 2.0 Gy = 10.0 Gy to 16.0 Gy, total dose 60.4 Gy to 66.4 Gy.

or Conventionaly fractionated radiotherapy of the breast 28 × 1.8 Gy = 50.4 Gy with simultaneous integrated boost to the tumor bed, total dose 28 × 0.3 Gy or 0.45 Gy= 8.4 Gy or 12,6 Gy, total dose 58,8 Gy to 63.0 Gy.

or Hypofractionated radiotherapy of the breast 16 × 2.66 Gy = 42.56 Gy followed by a tumor bed boost sequentially 5 to 8 × 2.0 Gy = 10.0 Gy to 16.0 Gy, total dose 52.56 Gy to 58.56 Gy.

Experimental Arm:

Hypofractionated radiotherapy of the breast 16 × 2.50 Gy with simultaneous integrated boost to the tumor bed, total dose within the boost volume 16 × 3.00 Gy.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically confirmed breast cancer operated by breast conserving surgery with clear margins independently of further risk factors (positive or high-risk negative lymph node status, estrogen- or progesterone receptor status, Her-2/neu status uPA/PAI-1 criteria) and postoperative systemic therapy (chemotherapy, endocrine, antibody or bisphosphonate therapy were permitted when indicated)
* Indication to adjuvant radiotherapy including boost radiotherapy
* Clearly identified primary tumor region preferably by radiopaque clips
* Primary wound healing after breast conserving therapy without signs of infection
* Age ≥ 18 years
* ECOG ≤ 2 Performance Status
* Written informed consent
* Compliance regarding treatment appointments and toxicity
* Linguistic and cognitive ability to understand the questionnaires

Exclusion Criteria:

* Patients operated by mastectomy
* No indication for boost radiation (e.g. status after IORT)
* double sided breast cancer
* Resection margins positive for disease or insufficient identification of the boost volume
* Indication for radiotherapy of the regional lymph nodes
* History of prior breast or thoracic radiotherapy
* Extended postoperative seroma at the beginning of radiotherapy
* Previously administered radiotherapy not allowing the required dose
* Pregnant or lactating patients and woman of child bearing potential, who lacked effective contraception
* treatment history of other cancer or participation in another clinical trial testing radiotherapy or drugs within 4 weeks of the start of treatment.
* Patients with serious, uncontrolled, physical or cerebrovascular disorders(e.g. myocardial infarction within the last 12 months) or neurologiy or psychiatric disorders thought to adversly affect treatment compliance

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2324 (Actual)
Dates: Start 2015-06-16 (Actual); Primary Completion 2019-01-08 (Actual); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 3 to 6 years
  any local or regional recurrence or distant metastasis or death

SECONDARY OUTCOMES:
Time to occurence of local recurrence | 3 to 6 years
  ipsilateral in-breast recurrence
Overall survival | 3 to 6 years
  death
Safety and side effects (Number of Patients with Adverse Events) | 3 to 6 years
  Number of Patients with Adverse Events
Acute and chronic toxicity (NCI-CTCAE) | 1 day, 7 days, end of radiation (last day of radiation and closing visite), 3 months, 6 months, 12 months, 18 months, 24 months, 30 months, 36 months, 42 months, 48 months, 54 months, 60 months, 66 months, 72 months
  All dimensions of NCI-CTCAE
Cosmetic results (NCI-CTCAE) | 1 day, end of radiation (last day of radiation and closing visite), 3 months, 12 months, 24 months, 36 months, 48 months, 60 months, 72 months
  NCI-CTCAE

CONTACTS AND LOCATIONS:
Overall Officials: Jürgen Dunst, MD, Study Chair — University Medical Center Schleswig-Holstein (UKSH)
Locations (88):
- Germany (88):
  - Gesundheitszentrum St.Marien Gmbh und Klinik für Strahlentherapie, Amberg
  - Medizinisches Versorgungszentrum Aue, Aue
  - Helios Kliniken Bad Saarow Klinik für Radioonkologie, Bad Saarow
  - HELIOS Klinikum Bad Saarow, Bad Saarow
  - Strahlentherapie Klinikum Bayreuth, Bayreuth
  - Medizinisches Versorgungs Zentrum Diagnostisch Therapeutisches Zentrum am Frankfurter Tor, Berlin
  - Strahlentherapie in Moabit /Praxis für Strahlentherapie, Berlin
  - Praxis für Radioonkologie und Strahlentherapie Berlin Südwest, Berlin
  - Ambulantes Gesundheitszentrum der Dr. med Maria Sternemann Charte -Universitätsmedizin Berlin, Berlin
  - Vivantes-Klinikum Berlin-Neukölln, Berlin
  - HELIOS Klinikum Berlin-Buch, Strahlentherapeutische Klinik, Berlin
  - Charite berlin (Virchow) Klinik für Strahlentherapie, Berlin
  - DRK Kliniken Berlin: Zentrum für Strahlentherapie MVZ pro patiente Westend, Berlin
  - MZV am HELIOS Klinikum Emil von Behring, Berlin
  - Gemeinschaftspraxis und Belegabteilung für Strahlentherapie, Bocholt
  - Ambulanz Bremen GMBH MVZ RadioOnkologie, Bremen
  - Zentrum für Strahlentherapie undRadioonkologie, Bremen
  - Krankenhaus Buchholz Abteilung für Strahlentherapie, Buchholz
  - Strahlentherapie Coesfeld, Coesfeld
  - Radiologie Strahlentherapie-Zweigpraxis vom MVZ Passau, Deggendorf
  - Praxis für Strahlentherapie Krankenhaus Dresden-Friedrichsstadt, Dresden
  - Malteser MVZ Duisburg-Süd, Duisburg
  - Universitätsklinikum Düsseldorf Klinik und Poliklinik für Strahlentherapie und Radioologische Onkologie, Düsseldorf
  - Gemeinschaftspraxis für Strahlentherapie und Radioonkologie, Elmshorn
  - MVZ Strahlentherapie Klinikum Esslingen GmbH, Esslingen am Neckar
  - Klinikum Frankfurt (Oder)Klinikum für Strahlentherapie Radioonkologie, Frankfurt (Oder)
  - Klinik für Strahlentherapie und Onkologie, Frankfurt/M
  - Strahlentherapie am Klinikum Fürth, Fürth
  - Strahlentherapiezentrum- Escher-Lippe(STZELL) und die Katholischen Kliniken-Emscher, Gelsenkirchen
  - Justus-Liebig Universität Gießen Strahlentherapie, Giessen
  - Praxis für Strahlentherapie Goch, Goch
  - Brustzentrum ALB FILS Kliniken GMBH, Göppingen
  - Ambulanzzentrum des UKE GmbH Bereich der Strahlentherapie, Hamburg
  - Radiologische Ambulanz Fachärzte für Radiologie,Nuklearmedizin und Strahlentherapie, Hamburg
  - Strahlenzentrum Hamburg, Hamburg
  - GSR Hameln, Hamelin
  - Gemeinschaftspraxis für Strahlentherapie und Radioonkologie / Hannover/Hildesheim/Hameln, Hanover
  - GSR Hannover Siloa, Hanover
  - Dr.med Jürgen Heide Facharzt für Strahlentherapie, Harburg
  - Gemeinschaftspraxis für Strahlentherapie und Radioonkologie(GSR), Hildesheim
  - Gemeinschaftspraxis für Strahlentherapie Hildesheim/Goslar, Hildesheim
  - Gemeinschaftspraxis für Strahlentherapie/Hildesheim/Goslar, Hildesheim
  - Strahlentherapie Hof, Hof
  - MVZ St. Vincent-Kliniken gAG, Karlsruhe
  - Praxis für Strahlentherapie am Universitätsklinikum Schleswig-Holstein, Kiel
  - Universitätsklinikum Schleswig-Holstein, Kiel
  - Universitätsklinikum Leibzig, Leipzig
  - Klinikum für Strahlentherapie - Klinikum Lippe, Lemgo
  - Klinikum Ludwigsburg Klinik für Radioonkologie, Ludwigsburg
  - Klinikum Lüneburg, Klinik für Strahlentherapie und Radioonkologie, Lüneburg
  - MVZ Prof.Dr.Uhlenbrock und Partner Strahlentherapie Lünen, Lünen
  - Klinik und Poliklinik für Radioonkologie und Strahlentherapie Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
  - Praxis für Strahlentherapie Mannheim, Mannheim
  - Universitätsklinikum Marburg Strahlentherapie und Radioonkologie, Marburg
  - Brustzentrum Helios Klinikum, Meiningen
  - MVZ Chariete Vivantes Gmbh Strahlentherapie, Mitte
  - Kliniken Maria Hilf Gmbh Klinik für Strahlentherapie, Mönchengladbach
  - Klinikum rechts der Isar, München
  - Klinik für Strahlentherapie- Radioonkologie, Münster
  - Praxis für Strahlentherapie und Radioonkologie am Clemenshospital, Münster
  - Strahlentherapie Neckarsulm, Neckarsulm
  - Dietrich Bonhoeffer Klinikum Neubrandenburg, Neubrandenburg
  - Praxis für Strahlentherapie Im Städtischen Klinikum Neunkirchen, Neunkirchen
  - Klinik für Strahlentherapie und Radioonkologie Pius-Hospital Oldenburg, Oldenburg
  - Zentrum für Strahlentherapie Rheine-Osnabrück, Osnabrück
  - MVZ Radio-LOG Schie in Altötting, Passau
  - Visiorad - Bereich Strahlentherapie, Pinneberg
  - Klinikum für Radioonkologie Klinikum Ernst von Bergmann, Potsdam
  - Krankenhaus Barmherzige Brüder Regensburg Medizinisches Versorgungszentrum, Regensburg
  - Überörtliche Gemeinschaftspraxis/Fachärzte für Strahlentherapie, Rheine
  - Kreiskliniken Esslingen Paracelsus Krankenhaus Ruit, Ruit
  - CaritasKlinikum Saarbrücken, Saarbrücken
  - XCare Praxis für Strahlentherapie, Saarlouis
  - MVZ Leopoldina Strahlentherapie, Schweinfurt
  - MVZ Leopoldina, Schweinfurt
  - Helios kliniken Schwerin GMBH, Schwerin
  - Johanniter Zentren für medizinische Versorgung in der Altmark GMBH, Stendal
  - Johanniter Zentrum für Medizinische Versorgung, Stendal
  - MVZ Klinikum Straubing GMBH Strahlentherapie, Straubing
  - MVZ-Uniklinik Tübingen gGmbH, Stuttgart
  - Praxis für Strahlentherapie Trier Ehrang, Trier
  - Universitätsklinikum Tübingen, Tübingen
  - Klinik für Strahlentherapie und Radioonkologie Universitätsklinikum Ulm, Ulm
  - Klinik für Strahlentherapie und Radioonkologie Schwarzwald-Baar -Klinikum, Villingen-Schwenningen
  - Praxis für Strahlentherapie und Radioonkologie am Krankenhaus Weilheim, Weilheim
  - Medizinisches Versorgungszentrum Wolfsburg GmbH, Wolfsberg
  - Universitätsklinikum Würzburg Klinik und Poliklinik für Strahlentherapie, Würzburg
  - Heinrich-Braun-Klinikum Zwickau, Zwickau

REFERENCES:
- [Background] Krug D, Vonthein R, Schreiber A, Boicev AD, Zimmer J, Laubach R, Weidner N, Dinges S, Hipp M, Schneider R, Weinstrauch E, Martin T, Horner-Rieber J, Olbrich D, Illen A, Hessler N, Konig IR, Dellas K, Dunst J. Impact of guideline changes on adoption of hypofractionation and breast cancer patient characteristics in the randomized controlled HYPOSIB trial. Strahlenther Onkol. 2021 Sep;197(9):802-811. doi: 10.1007/s00066-020-01730-9. Epub 2020 Dec 15. PMID 33320286